CLINICAL TRIAL: NCT06417502
Title: Observational Study of Pediatric Rheumatic and Immunologic Diseases in China: The CAPRID Registry
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other); Central South University (Other); Beijing Children's Hospital (Other); Shenzhen Children's Hospital (Other Government); Children's Hospital of Nanjing Medical University (Other); The University of Hong Kong (Other); Zhejiang University (Other); Third Hospital of Peking University (Unknown)
Responsible Party: Principal Investigator, Hongmei Song, MD, Peking Union Medical College Hospital
Other Study IDs: JS-3362D; 2021YFC2702000 (Other Grant/Funding Number: National Key R&D Program of China)
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Autoimmune Diseases; Autoinflammatory Diseases
Keywords: Systemic Lupus Erythematosus; Juvenile Idiopathic Arthritis; Vasculitis; Juvenile Dermatomyositis; Sjogren's disease; Autoimmune; Autoinflammatory Disease; Scleroderma
MeSH Terms: conditions — Autoimmune Diseases; Lupus Erythematosus, Systemic; Arthritis, Juvenile; Vasculitis; Dermatomyositis; Sjogren's Syndrome; Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational, multi-center, longitudinal registry study for Chinese pediatric patients with rheumatic and immunologic diseases.

DETAILED DESCRIPTION:
Pediatric rheumatic and immunologic diseases severely impact the health of children and adolescents. Chinese Alliance of Pediatric Rheumatic & Immunologic Diseases (CAPRID) was founded in 2022 to form a national collaboration for high-quality data-driven multi-center pediatric rheumatology and immunology research in China. The CAPRID Registry is an observational, multi-center, longitudinal registry for Chinese pediatric patients with rheumatic and immunologic diseases to explore the clinical phenotypes, diagnoses, complications, real-world drug safety, therapeutic efficacy, adverse events, critical illness and outcomes of Chinese pediatric patients with rheumatic and immunologic diseases.

Hospital-based databases are established and standardized with Observational Medical Outcomes Partnership (OMOP) Common Data Model (CDM) for routine data collection. A web-based registry website is established with standardized electronic case report forms to register patients from CAPRID centers. A mobile application is created to allow long-term follow up and patient-reported outcome collection. The data captured in this registry reflects a "real world" situation with no intervention done outside the routine clinical practice. Treatment plans are determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age <= 18 years old
* Diagnosed with rheumatic and immunologic diseases (including diffuse connective tissue diseases, arthritis, vasculitis, inborn errors of immunity)
* Diagnosed and Treated in China

Exclusion Criteria:

* Disagreement of involving in this study by the patient or his/her family.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Chinese children with pediatric rheumatic and immunologic diseases enrolled from CAPRID centers.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Enrolled Patients | up to 10 years
  Total number of patients with pediatric rheumatic and immunologic diseases enrolled in the registry

SECONDARY OUTCOMES:
Physician Global Assessment | up to 10 years
  Visual Analog Score measurement of disease activity by physicians. The minimum value is 0 and the maximum is 10.
Patient or Parent Global Assessment | up to 10 years
  Visual Analog Score measurement of disease activity by patient's parent or patient him or her self (above 8 years old). The minimum value is 0 and the maximum is 10.
Proportion of Participants with Clinically Inactive Disease | up to 10 years
  Defined by normal disease activity indexes (if available) and normal inflammatory markers (erythrocyte sedimentation rate and C-reactive protein).
  Disease activity indexes include Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) for systemic lupus erythematosus; Juvenile Arthritis Disease Activity Score (JADAS)-27 for juvenile idiopathic arthritis, Pediatric Vasculitis Activity Score (PVAS) for vasculitis; Manual Muscle Testing(MMT)8, Childhood Myositis Assessment Scale (CMAS) for juvenile dermatomyositis, Sjögren's syndrome disease activity index (ESSDAI) for Sjögren's syndrome, Modified Rodnan Skin Score for scleroderma.
Childhood Health Assessment Questionnaire (CHAQ) | up to 10 years
  Composite measure of functional disability, score from 0 (no disability) to 3 (severe disability)

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Song, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (9):
- China (9):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Third Hospital of Peking University, Beijing, Beijing Municipality
  - Chidren's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - The University of Hong Kong Shenzhen Institute of Research and Innovation (HKU-SIRI), Shenzhen, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

REFERENCES:
- See also: The Official Website for Chinese Alliance of Pediatric Rheumatic & Immunologic Diseases (CAPRID) — https://caprid.pumch.cn